CLINICAL TRIAL: NCT05783557
Title: A Randomized, Double-blind, Active-compared Phase Ш Clinical Trial to Evaluate Clevidipine Butyrate Injectable Emulsion in the Treatment of Hypertensive Emergency and Sub-emergency
Brief Title: A Study of Clevidipine Butyrate Injectable Emulsion in the Treatment of Hypertensive Emergency and Sub-emergency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC1902-002
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hypertensive Emergency
MeSH Terms: conditions — Hypertensive Crisis | interventions — clevidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group
  Interventions: Drug: Clevidipine Butyrate Injectable Emulsion
- Active-compared Group (Active Comparator): Active-compared Group
  Interventions: Drug: Cleviprex®

INTERVENTIONS:
Drug: Clevidipine Butyrate Injectable Emulsion — intravenous injection
  Other Names: HC1902
  Arms: Experimental Group
Drug: Cleviprex® — intravenous injection
  Other Names: Clevidipine Butyrate Injectable Emulsion
  Arms: Active-compared Group

SUMMARY:
A randomized, double-blind, active-compared phase Ш clinical trial to evaluate clevidipine butyrate injectable emulsion in the treatment of Hypertensive Emergency and Sub-emergency.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, active-compared Phase III clinical study to evaluate the efficacy and safety of clevidipine butyrate injectable emulsion in the treatment of Hypertensive Emergency and Sub-emergency. The Cleviprex® will be chosen as the positive controlled medicine with the same usage of the test drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years-old and ≤75 years-old, regardless of gender;
2. Patients with hypertensive emergency and sub-emergency requiring a rapid intravenous blood-pressure control: patients with SBP > 180 mmHg and/or DBP > 120 mmHg (requiring twice consecutive blood pressure measurements, 10 to 15 min apart), with or without target organ damage;
3. A potentially fertile patient is willing and required to use reliable contraceptive methods throughout the study period and for at least 3 months after initiation of test drug to avoid pregnancy in the female patient or in the male patient's partner;
4. Able to understand informed consent, participate in the experiment voluntarily and sign informed consent.

Exclusion Criteria:

1. Antihypertensive drugs have been used within 2 hours before the administration of test drugs;
2. Patients with life-threatening clinical manifestations, such as malignant arrhythmias, respiratory failure, and severe disturbance of consciousness;
3. Patients with confirmed or suspected severe aortic stenosis or aortic dissection at screening time;
4. Patients with obstructive hypertrophic cardiomyopathy and systolic heart failure at screening time;
5. Patients with acute coronary syndrome at screening or myocardial infarction within 1 month before screening;
6. Patients with acute stroke within 1 month before screening;
7. Patients with clear history of secondary hypertension;
8. Patients with lipid metabolism defects;
9. Patients with a known history of liver failure or cirrhosis;
10. Patients with chronic kidney disease (CKD) stage 5, requiring long-term regular dialysis treatment;
11. Patients who are allergic to the test drug or its ingredients, or who are intolerant to calcium channel blockers, or who are allergic to soy, soy products, eggs and egg products;
12. Patients with mental illness, mental disorder and other disorders who cannot communicate properly;
13. A history of drug abuse, drug use, or alcohol dependence;
14. Female patients who are pregnant or lactating;
15. Patients who have participated in other interventional clinical trials within 3 months prior to screening;
16. Patients who are judged by the investigators to be ineligible for this study for other factors, such as patients who could not receive intravenous infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients whose SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30 minutes of administration | 30 minutes
  Proportion of patients whose SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30 minutes of administration

SECONDARY OUTCOMES:
The time for the first SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30minutes min of within 30 minutes of administration | 30 minutes
  The time for the first SBP fell within the target range (SBP decreased by ≥15% and ≤25% from baseline) within 30 minutes of within 30 minutes of administration
AUC above the upper limit of the target range and below the lower limit of the target range within 1 hour of administration | 1 hour
  AUC above the upper limit of the target range and below the lower limit of the target range within 1 hour of administration
Proportion of patients successfully converted to oral antihypertensive therapy within 6 hours of discontinuation | 6 hours
  Proportion of patients successfully converted to oral antihypertensive therapy within 6 hours of discontinuation
Change of heart rate from baseline within 30 min of administration | 30 minutes
  Change of heart rate from baseline within 30 min of administration
Incidence of adverse events (AEs) | Throughout the study period, within 72 hours
  Incidence of adverse events (AEs)
Total dosage of clevidipine butyrate injectable emulsion | Throughout the study period, within 72 hours
  Total dosage of clevidipine butyrate injectable emulsion

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Principal Investigator — Beijing Anzhen Hosipital, Capital Medical University